CLINICAL TRIAL: NCT04887220
Title: Persistent Pain and Its Impact on Quality of Life at 3, 6 and 12 Months in COVID-19 Patients Who Have Required Critical Care
Brief Title: Persistent Pain and Its Impact on Quality of Life COVID-19 Patients That Required Critical Care
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-COV-2020-63
Record Dates: First submitted 2021-01-21; First posted 2021-05-14 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Chronic Pain; Post ICU Syndrome; Quality of Life
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 infection produces thousands of hospital admissions in a very short period of time, including critical care patients. It is expected that those who survive a severe spectrum of the disease, will present some degree of health decline in the medium and long term, becoming chronic patients.

Post-intensive care syndrome (PICS) was described by the Society of Critical Care Medicine (SCCM) as a new altered or worsening of physical, cognitive, or mental condition due to critical illness and persisting after hospitalization, including pain. Also, clinical features of infection include different types of pain, and if this pain persists, it can turn into a chronic condition. Chronic pain is a currently recognized disease, but under-treated in many cases, generating a significant deterioration in the quality of life of this patient. It is vitally important to generate early care circuits to detect and treat those expected complications, such as chronic pain in these patients. The objective of this study is to estimate the level of persistent pain and its impact on health-related quality of life after admission to an intensive care unit in patients who suffered this infection.

DETAILED DESCRIPTION:
The presence of persistent pain and impaired quality of life in COVID19 patients who have required intensive care can affect up to a total of 50% of patients.

Main objective Estimate the level of persistent pain and health-related quality of life after admission one in intensive care unit in COVID-19 patients, a new disease that has been accompanied by great health, social and economic involvement from which we do not know the long-term consequences in this patient cohort.

Secondary goals

* Assessing patient's characteristics before ICU admissión; the prevalence of painkillers use, including opioids, history of previous pain, and comorbidities. Find relationships between these characteristics and the development of chronic pain.
* Determine if some ICU treatments and patient's characteristics may contribute to persistent pain in COVID-19 survivors ( number of prone therapies, thromboembolic complications, and medication for sedate used)
* Determine the quality of life using the SF-12 test.
* Determine pain characteristics using the ID-PAIN test.
* Determine the scale of anxiety and depression using the HADs test.

ELIGIBILITY:
Inclusion Criteria:

* Post ICU COVID 19 Survivor
* Adult 18 year or older, who gives its approval to participate

Exclusion Criteria:

* Refusal to participate
* Neurological or physical secuale, disabled to answer a questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults survivors after critical state of COVID 19, who requires critical care.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
VAS scale value | 1 year
  Chronic pain in PostICU COVID19 survivors, measured by VAS scale from Brief Pain Inventory Questionnaire

SECONDARY OUTCOMES:
Quality of life score | 1 year
  Quality of life assessment by SF-12 questionnarie, of ICU survivors after 12 months of ICU discharge
ID Pain test value | 1 year
  Pain characteristics of ICU COVID 19 survivors, using ID PAIN test for presence of neuropathic pain
HAD scale value | 1 year
  Level of anxiety and/or depression in post ICU survivors of COVID 19 at 12 months after discharge, using HAD questionnarie

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided